CLINICAL TRIAL: NCT05460117
Title: Elastography and Thermography Plantar Fasciopathy Assessment After Radiofrequency Stimulation in a Sporty Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Daniel Aguilar Nunez, Clinical Professor, University of Malaga, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DAN15
Record Dates: First submitted 2022-06-26; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fascia; Contracture
MeSH Terms: conditions — Contracture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency stimulus on the dominant PLANTAR FASCIOPATHY (Experimental): 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus on the dominant Plantar fasciopathy
  Interventions: Device: Radiofrecuency

INTERVENTIONS:
Device: Radiofrecuency — he use of 448kilohertz capacitive resistive monopolar radiofrequency as the focus of the treatment looking for improve the quality of the tissue is still to be explored.

SUMMARY:
448kilohertz capacitive resistive monopolar radiofrequency is a novel technique in physiotherapy and its usefulness and clinical relevance is still to be investigated at both clinical practice and also in performance. Current studies show promising results in different musculoskeletal disorders, however there no studies in the assessment of quality soft tissue in sporty population after the used of this technique.

DETAILED DESCRIPTION:
Plantar Fasciopathy pain is is one of the most common musculoskeletal disorders, presenting a high prevalence in primary care centers and sport populations. Many factors have been proposed as the cause of pain, however there are no studies analysing possibilities of preventing foot injuries by using a radiofrequency stimulus.

The use of 448kilohertz capacitive resistive monopolar radiofrequency as the focus of the treatment looking for improve the quality of the tissue is still to be explored.

The hypothesis of the present project is that focus treatments on 448kilohertz capacitive resistive monopolar radiofrequency on the shoulder will produce better outcomes in terms of ultrasound assessment measured by quantified elastography, and this will decreased the possibilities of get injured.

All interventions will be developed by the same examiner, who is a physiotherapist with 6 years of clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years --Sporty people with at least 3 days of training per week and presenting an upper limb dominance

Exclusion Criteria:

* Suffer from any painful shoulder condition.
* History of significant shoulder trauma, such as fracture or ultrasonography
* Clinically suspected partial thickness cuff tear, following the classification of Wiener and Seitz.
* Recent shoulder dislocation in the past two years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-12 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in plantar fasciopathy measured by quantified elastography.imaging at 3 months [ Time Frame: Time Frame: time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)]. Changes in tendinous thickness | 9 months
  The elastography is obtained when the anatomic image on grayscale ultrasound overlaps parametric color image that expresses the rate of deformity of the tissues, soft tissues tend to develop greater deformity and tissue deformity have lower rigidity.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Ana Gonzalez, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided